CLINICAL TRIAL: NCT01388478
Title: Safety/Tolerability and Effects on Cognitive Impairment, Impaired Cerebral Cortical Metabolism and Oxidative Stress of R(+)Pramipexole Administered to Subjects With Early Alzheimer's Disease
Brief Title: Safety Study of R(+)Pramipexole to Treat Early Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of Kansas (Other); Alzheimer's Drug Discovery Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCU-KU-ADDF-2011; 20101202 (Other Grant/Funding Number: Alzheimer's Drug Discovery Foundation)
Record Dates: First submitted 2011-06-30; First posted 2011-07-06 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Alzheimer's Disease
Keywords: Safety; Tolerability; R(+)Pramipexole; Alzheimer's
MeSH Terms: conditions — Alzheimer Disease | interventions — Dexpramipexole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R(+)pramipexole (Experimental): Each study participant will be given the active study drug, R-pramipexole. There is no placebo arm.
  Interventions: Drug: R-pramipexole

INTERVENTIONS:
Drug: R-pramipexole — R-pramipexole will be taken as a liquid and start at one teaspoon (5 ml) twice a day for a total dose of 100 mg/day. After 4 weeks, the dose will double (two teaspoons twice a day, or a total of 200mg/day). Four weeks later the dose will be increased again to 2 1/2 teaspoons twice a day (total of 300mg/day) where it will remain for the remaining 16 weeks of study treatment. Prior to each increase, participants and their study partners will be interviewed regarding any possible side effects or problems. These findings will be discussed with the physician prior to increasing the study drug dose. The dose will only increase if the participant is not having side effects.
  Other Names: Dexpramipexole

SUMMARY:
By doing this study, researchers will examine the safety and tolerability of R-pramipexole in participants with Alzheimer's disease. This study will also examine the body and brain's response to the study drug by measuring the amount of injury to the cells (oxidative stress) in the blood and spinal fluid and brain imaging before and after treatment.

DETAILED DESCRIPTION:
Subjects will be recruited from the Univ of Kansas Alzheimer's Center and will provide informed consent about participating.

R(+)-pramipexole will be provided as Good Manufacturing Practice powder and taken as a liquid and start at one teaspoon (5 ml) twice a day for a total dose of 100 mg/day. After 4 weeks, the dose will double (two teaspoons twice a day, or a total of 200mg/day). Four weeks later the dose will be increased again to 2 1/2 teaspoons twice a day (total of 300mg/day) where it will remain for the remaining 16 weeks of study treatment. Prior to each increase, participants and their study partners will be interviewed regarding any possible side effects or problems. These findings will be discussed with Dr. Burns prior to increasing the study drug dose. The dose will only increase if the participant is not having side effects.

Primary Outcome Measure:

1.Number of Patients with Adverse Events [Time Frame: Every 2 months] [Safety Issue: Yes]

Labwork will be performed every two months. There will be frequent contact with subjects to assess for adverse events.

Secondary Outcome Measures:

Reduction of Oxidative Stress [Time Frame: Baseline and at 24 weeks after taking study drug] [Safety Issue: No]

A lumbar puncture (spinal tap) will be performed to collect cerebral spinal fluid, which will be assayed for isoprostane levels before and after treatment.

Changes in cerebral glucose metabolism [Time Frame: Baseline and at 24 weeks after taking drug] [Safety Issue: No]

Positron Emission Tomography Scan will be performed. Changes in cerebral glucose metabolism as a proxy for mitochondrial respiration will be assayed at baseline and 24 weeks. Correlations will be sought with assays of oxidative stress reduction to see if greater reductions in brain oxidative stress are reflected in elevations of cortical 2-fluorodeoxyglucose.

Effects on Cognitive Performance [Time Frame: Baseline and then 6 months thereafter] [Safety Issue: Yes]

Quantitative assessment of cognitive status will be taken at baseline and at end of 6 month dosing period.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided by the participant or the participant's legally acceptable representative
* Age 55 years or older
* Possible/probable Alzheimer's Disease (AD)
* Community dwelling with a caregiver able and willing to accompany the participant on all visits, if necessary. Caregiver must visit with the subject >5 times per week.
* Rosen Modified Hachinski score of 4 or less
* Imaging Study (CT or MRI) compatible with AD or age-related changes (absence of significant abnormalities that may explain cognitive decline, such as multiple lacunar infarcts or a single prior infarct >1 cubic cm, microhemorrhages or evidence of a prior hemorrhage > 1 cubic cm, evidence of cerebral contusion encephalomalacia, aneurysm, vascular malformation, or space occupying lesion such as an arachnoid cyst or brain tumor).
* Adequate visual and auditory abilities to perform all aspects of the cognitive and functional assessments

Exclusion Criteria:

* Significant neurological disease, other than AD, that may affect cognition
* Current clinically-significant systemic illness that is likely to result in deterioration of the patient's condition or affect the patient's safety during the study.
* History of clinically-evident stroke
* Clinically-significant infection within the last 30 days
* Myocardial infarction or symptoms of active coronary artery disease (e.g., angina) in the last two years.
* Uncontrolled hypertension within the last 6 months.
* History of cancer within the last 5 years (except non-metastatic basal or squamous cell carcinoma)
* History of drug or alcohol abuse as defined by DSM-IV criteria within the last 2 years
* Insulin dependent diabetes mellitus
* Significant pain or musculoskeletal disorder that would prohibit participation in metabolic testing

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P. Bennett, MD, PhD, Principal Investigator — Virginia Commonwealth University; Jeffrey M Burns, MD, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | R(+)Pramipexole
Started | 20
Completed | 15
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | R(+)Pramipexole
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events
Description: Labwork will be performed every two months. There will be frequent contact with subjects to assess for adverse events.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | R(+)Pramipexole
Number analyzed (Participants) | 20
Participants | 18

2. Other Pre Specified Outcome: Effects on Cognitive Performance
Description: Quantitative assessment of cognitive status will be taken at baseline and at end of 6 month dosing period.
Time Frame: Baseline and then 6 months thereafter
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Changes in Cerebral Glucose Metabolism
Description: PET Scan will be performed. Changes in cerebral glucose metabolism as a proxy for mitochondrial respiration will be assayed at baseline and 24 weeks. Correlations will be sought with assays of oxidative stress reduction to see if greater reductions in brain oxidative stress are reflected in elevations of cortical 2-FDG.
Time Frame: Baseline and at 24 weeks after taking drug
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Reduction of Oxidative Stress
Description: A lumbar puncture (spinal tap) will be performed to collect cerebral spinal fluid, which will be assayed for isoprostane levels before and after treatment.
Time Frame: Baseline and at 24 weeks after taking study drug
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | R(+)Pramipexole
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 18/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R(+)Pramipexole (N=20)
Agitation/irritability (Psychiatric disorders) | 2 (2)
Tooth problems (General disorders) | 2 (2)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cold symptoms (Infections and infestations) | 1 (1)
Confabulations (Nervous system disorders) | 1 (1)
Contusion (Nervous system disorders) | 2 (2)
Coughing (General disorders) | 1 (1)
Decreased appetite (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dreaming (Psychiatric disorders) | 2 (2)
Falls (Nervous system disorders) | 5 (5)
Hallucinations (Nervous system disorders) | 2 (3)
Increased confusion (Nervous system disorders) | 3 (5)
Increased depression (Psychiatric disorders) | 1 (1)
Increased libido (Endocrine disorders) | 3 (3)
Injury to urethra (Renal and urinary disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3)
Laceration (Skin and subcutaneous tissue disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Nausea or vomiting (Gastrointestinal disorders) | 4 (4)
Sensation in throat (General disorders) | 1 (1)
Sinus issues (General disorders) | 2 (2)
Sleep disturbance (Nervous system disorders) | 4 (5)
Somnolence (Nervous system disorders) | 1 (1)
Sweating (General disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-02-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT01388478/Prot_SAP_000.pdf